CLINICAL TRIAL: NCT02706665
Title: Modelling Pharmacokinetic/Pharmacodynamic of Propofol Based on PSI Values From the SEDline®
Brief Title: Monitoring of Hypnosis State During General Anesthesia With Propofol by Patient State Index From SEDLine®
Status: Completed | Type: Observational
Sponsor: Hospital Universitario de Canarias (Other)
Collaborators: Masimo Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 2013_10
Record Dates: First submitted 2016-03-07; First posted 2016-03-11 (Estimated); Last update posted 2019-10-17 (Actual); Status verified 2016-03

CONDITIONS: Hypnotic Effect
Keywords: Anesthetics; Propofol; Electroencephalography; SEDline monitor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: SEDline monitor — The SEDline monitor gives us the Patient State Index (PSI), a dimensionless number within a range of 0 to100.

SUMMARY:
The purpose of this study is the evaluation of possible relationships and correlation between PSI values obtained from the SEDLine® monitor and the infusion rate of propofol during general anesthesia.

DETAILED DESCRIPTION:
Introduction:

There is a large intra-and interindividual variability in the effect of propofol. To deal with this problem, a real-time monitoring and therefore a more accurate titration of anesthetic agents is proposed. Brain function monitors based on a processed analysis of EEG (Electroencephalogram) can help to control pharmacodynamic effects of hypnotic agents. PSI values provide a measurement of the hypnotic effect of propofol. It will be observed an inverse correlation between the propofol infusion rate and the PSI value.

Objectives:

To design a computer program to record simultaneously the propofol infusion rate, PSI and Electromyogram (EMG).

To study the correlation between PSI values obtained from the SEDLine® monitor and the infusion rate of propofol during general anesthesia.

To obtain a mathematical model of the system from data recorded with different identification techniques.

Methods:

A group of patients scheduled for surgery under a standard total intravenous anesthesia (TIVA) with propofol and remifentanil will be recruited. The hypnotic effect of propofol will be monitored with the PSI from a SEDline monitor continuously. All anesthetic doses and their changes fall within conventional dosing.

The procedure for recording data and obtaining the pharmacokinetics/pharmacodynamics (PK / PD) model will be connecting a SEDLine® monitor to a laptop with an original program developed by members of our team. The program automatically stores the infusion rate of propofol (mg/kg/h) and the simultaneous values of PSI and frontal EMG. Graphics and data collected will be explored with various systems of techniques for pattern recognition in order to get the best fit to define a mathematical model of the dose of propofol and PSI values. A subsequent computer analysis with MATLAB® will estimate the correlation between the infusion of propofol infusion rate and PSI values.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists classification of I, II, or III
* Patient signed an informed consent

Exclusion Criteria:

* Patients with prior neurological disease, epilepsy or stroke.
* Patients who are receiving drug therapy that may alter processed EEG monitoring and decrease the PSI accuracy.
* American Society of Anesthesiologists classification IV or higher

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inpatients undergoing a surgery procedure with general anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2015-12; Primary Completion 2016-06 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
EEG processed will be measured by non invasive adhesive electrodes on the skin of the forehead's patient. A disposable sensor connected with a SEDLine provides de PSI index | During general anaesthesia in the operating room for a scheduled surgery.
  The values from the SEDLine ® monitor inversely correlate with the rate of infusion of propofol. Changes in that velocity correspond to changes in the effect site (CNS) and are related to the PSI values displayed in the monitor.

SECONDARY OUTCOMES:
Time from discontinuation of intravenous agents to open eyes to order | In the operation room at the end of surgery
  It will be measured with a chronometer

CONTACTS AND LOCATIONS:
Overall Officials: Jose Antonio Reboso Morales, MD, PhD, Principal Investigator — Hospital Universitario de Canarias
Locations (1):
- Hospital Universitario de Canarias, San Cristóbal de La Laguna, Santa Cruz De Tenerife, Spain